CLINICAL TRIAL: NCT06818773
Title: Efficacy and Safety Study of Inetetamab Combined with Chemotherapy ± PD-1/PD-L1 Inhibitor As First-Line Treatment for HER2-Positive Advanced Biliary Tract Cancer
Brief Title: Inetetamab Plus Chemotherapy ± PD-1/PD-L1 in HER2+ Advanced Biliary Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Dean of the Clinical Research Institute, Director of the Department, Eastern Hepatobiliary Surgery Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-FB-SC-09-V1.3
Record Dates: First submitted 2024-12-29; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Biliary Tract Cancer; HER2 Positive
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- inetetamab+ Gemcitabine + Cisplatin ± PD-1/PD-L1 Inhibitor (Experimental)
  Interventions: Drug: Inetetamab + Gemcitabine + Cisplatin ± PD-1/PD-L1 inhibitor

INTERVENTIONS:
Drug: Inetetamab + Gemcitabine + Cisplatin ± PD-1/PD-L1 inhibitor — A 21-day cycle is used, with the initial dose of inetuximab at 8 mg/kg (IV), followed by 6 mg/kg (IV) on Day 1 of each subsequent cycle. Gemcitabine (1000 mg/m²) + cisplatin (25 mg/m²) are administered in combination on Day 1 and Day 8 of each cycle. The appropriate PD-1/PD-L1 inhibitor will be selected by the investigator based on the patient's specific condition, and its administration will strictly follow the dosing instructions provided in the relevant drug's package insert.

SUMMARY:
To evaluate the efficacy and safety of inetetamab in combination with chemotherapy ± immunotherapy as a first-line treatment for HER2-positive advanced biliary tract cancer, providing theoretical evidence and practical guidance for further optimizing treatment regimens and improving therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years;
* Histologically confirmed HER2-positive metastatic biliary tract cancer;
* ECOG performance status of 0 to 1;
* No prior treatment with anti-HER2 therapies;
* Patients have not received any systemic anticancer treatment in the recurrent/metastatic setting;
* Patients who have experienced disease recurrence more than 6 months after curative surgery; if adjuvant therapy (chemotherapy and/or radiotherapy) was received post-surgery, patients must have had recurrence more than 6 months after completion of adjuvant therapy;
* Presence of at least one measurable lesion;
* Adequate function of major organs as defined by the following criteria;
* Estimated survival of ≥3 months;
* Voluntary participation in this study, signing of the informed consent form, good compliance, and willingness to cooperate with follow-up.

Exclusion Criteria:

* Known allergy or contraindication to any component of the study drugs;
* Previous treatment with anti-HER2 therapies;
* Prior use of immunotherapy;
* Use of immunosuppressive agents within 14 days before the first dose, except:

Intranasal, inhaled, topical steroids, or local injections (e.g., intra-articular) Systemic corticosteroids ≤10 mg/day prednisone or equivalent Steroids for hypersensitivity reactions (e.g., premedication for CT scans)

* Known active central nervous system metastases or carcinomatous meningitis;
* Other malignancies within 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell skin cancer;
* Major surgery or significant trauma within 4 weeks before randomization, or planned major surgery;
* Severe cardiac disease;
* Resting dyspnea due to tumor progression or comorbidities, or requiring supplemental oxygen;
* Neuropathy ≥ Grade I per NCI criteria;
* Active interstitial lung disease (ILD) or pulmonary disease requiring bronchodilators;
* History of immunodeficiency;
* Participation in another drug trial within 4 weeks before screening;
* Pregnant or breastfeeding women, or women of childbearing potential with a positive pregnancy test at screening; unwillingness to use effective contraception during and for 6 months after the study;
* Any serious concomitant illness or conditions that may interfere with the planned therapy or render participation unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 months

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 12 months
Disease Control Rate (DCR) | 12 months
Overall Survival (OS) | 24 months
Quality of Life Questionnaire-Core 30（QLQ-C30） | 24months
Adverse Event（AE） | 24 months